CLINICAL TRIAL: NCT00224419
Title: Testing Pharmacological Therapies for Pregnant Smokers
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: was terminated due to meeting a priori stopping rule set by DSMB
Sponsor: Duke University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Kathryn Pollak, PhD, Duke University Department of Community and Family Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00007724; Duke University IRB #2865; CA89053 (Other: DUMC)
Record Dates: First submitted 2005-09-21; First posted 2005-09-23 (Estimated); Last update posted 2014-07-21 (Estimated); Status verified 2009-04

CONDITIONS: Smoking; Pregnancy
Keywords: Smoking cessation; Pregnancy; Nicotine replacement therapy; Motivational interviewing
MeSH Terms: conditions — Smoking; Smoking Cessation | interventions — Motivational Interviewing; Nicotine; Transdermal Patch; Chewing Gum; Nicotine Replacement Therapy; Nicotine Chewing Gum

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 - CBT Counseling (Active Comparator): Participants in this arm received a tailored CBT (TCBT) intervention that included: a written self-help guide, feedback about the importance of reducing nicotine exposure to the fetus, 5 face to face and 1 telephone counseling session.
  Interventions: Behavioral: Motivational interviewing for smoking cessation; Behavioral: Cognitive behaviors therapy
- 2 - Counseling + NRT (Experimental): Women in this arm received the TCBT described in Arm 1, plus their choice of NRT. To minimize fetal exposure to nicotine for women in the TCBT+NRT arm, the dose of NRT are customized to the woman's current level of smoking. Women who smoke 5-10 cigarettes a day will be given the 14 mg patch or instructed to use one 2 mg lozenge or 2 mg piece of gum to replace each cigarette she usually smokes per day. Those who smoke 11 cigarettes or more per day will be given the 21 mg patch or instructed to use no more than one lozenge (2 mg) or piece of gum (2 mg) to replace each cigarette she usually smokes per day, not to exceed 15 lozenges or pieces of gum per day.
  Interventions: Behavioral: Motivational interviewing for smoking cessation; Drug: CBT + NRT

INTERVENTIONS:
Behavioral: Motivational interviewing for smoking cessation — All participants received a tailored CBT (TCBT) intervention that included: a written self-help guide, info about the importance of reducing nicotine exposure to the fetus, 5 face to face and 1 telephone counseling session. Women in the TCBT + NRT arm were guided through a process of deciding on nicotine gum, lozenge or patch. To minimize fetal exposure, the dose of NRT was customized to the woman's current level of smoking. Women who smoked 5-10 cigarettes a day were given the 14 mg patch or instructed to use one 2 mg lozenge or 2 mg piece of gum to replace each cigarette she usually smoked per day. Those who smoked 11 cigarettes or more per day were given the 21 mg patch or instructed to use no more than one lozenge (2 mg) or piece of gum (2 mg) to replace each cigarette she usually smoked per day, not to exceed 15 lozenges or pieces of gum per day.
  Other Names: Nicoderm CQ (patch); Nicorertte (gum); Commit (lozenge)
Behavioral: Cognitive behaviors therapy — 6 counseling sessions delivered over the phone or in person
  Arms: 1 - CBT Counseling
Drug: CBT + NRT — Includes CBT from arm 1 plus choice of NRT (lozenge, gum, or patch) tailored to smoking amount
  Other Names: Nicoderm CQ (patch); Nicorette (gum); Commit (lozenge)
  Arms: 2 - Counseling + NRT

SUMMARY:
Nicotine dependence has not been sufficiently addressed in current state-of-the-science cessation interventions for pregnant smokers. The weight of the evidence from the general population of smokers suggests that nicotine replacement therapies may be beneficial cessation aids for pregnant smokers who are unable to stop smoking. The tremendous potential of these therapies for promoting smoking cessation among pregnant women creates a pressing need for decision tools and protocols to encourage treatment adherence that is essential for rigorous evaluation of the effectiveness of OTC NRT when provided as part of prenatal care. The results of this research could be directly translated to the improvement of obstetrical care providers' clinical practices. Medically supervised use of OTC NRT by pregnant smokers is an alternative to continued smoking that has the potential to substantially increase rates of smoking cessation during pregnancy.

DETAILED DESCRIPTION:
The proposed five-year study is designed to evaluate the effectiveness of providing over-the-counter (OTC) nicotine replacement therapy, choice of gum, lozenge or patch, (NRT) to promote prepartum smoking cessation. Proposed is a two-arm design. Eligible pregnant women (N=300) will be randomized to either: Arm 1, Tailored Cognitive Behavioral Treatment (TCBT, n=100) that provides women with customized risk information about smoking and nicotine, the potential harms to the fetus and encouragement of appropriate behavioral skills building; or Arm 2, TCBT + NRT - the tailored intervention incorporating NRT information plus choice of patch or gum (n=200). The intervention will include 5 face-to-face contacts as part of prenatal visits and 1 telephone counseling session. Primary outcome measures will be biochemically validated 7-day prevalent abstinence rates at the 19-27th and 29-37th week of pregnancy. Secondary outcomes will include 7-day prevalent abstinence rates at 12 weeks postpartum, serious quit attempts, compliance with NRT, and use of materials. Saliva cotinine will be measured among all women at baseline, the 27-35th week of pregnancy, and 12 weeks postpartum. The significance of this project is that it relies on transdisciplinary collaborations to extend the science in nicotine replacement therapies to a population that could derive substantial health benefits. Moreover, the study results have immediate potential to inform clinical recommendations for integrating nicotine replacement into prenatal care.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age
* Be between 13 and 25 weeks of pregnancy
* Be receiving prenatal care at one of the participating clinics
* Have smoked at least 100 cigarettes in their lifetime
* Be currently smoking and have smoked at least 5 cigarettes per day in the past 7 days
* Speak and write English

Exclusion Criteria:

* Evidence of cognitive or mental health problems
* Evidence of possible drug or alcohol addiction
* Documented history in medical chart of mental retardation, significant chronic or recurrent psychiatric disorder such as schizophrenia or severe depression, history of cardiac arrhythmias, history of myocardial infarction within the past 6 months, history of previous pregnancy with congenital anomaly,family history of congenital anomalies
* Complications of pregnancy during the current pregnancy, including: threatened miscarriage, congenital anomalies, unexplained vaginal bleeding, pelvic or abdominal surgical procedures, deep venous thrombosis, malignancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2003-06; Primary Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Biochemically-validated smoking cessation | middle and late pregnancy

SECONDARY OUTCOMES:
Biochemically-validated smoking cessation | 3 months postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Evan Myers, MD, MPH, Principal Investigator — Duke University
Locations (2):
- United States (2):
  - Duke University Medical Center, Durham, North Carolina
  - Womack Army Medical Center, Fayetteville, North Carolina

REFERENCES:
- [Background] Pletsch PK, Pollak KI, Peterson BL, Park J, Oncken CA, Swamy GK, Lyna P. Olfactory and gustatory sensory changes to tobacco smoke in pregnant smokers. Res Nurs Health. 2008 Feb;31(1):31-41. doi: 10.1002/nur.20229. PMID 18161772
- [Background] Pollak KI, Oncken CA, Lipkus IM, Peterson BL, Swamy GK, Pletsch PK, Lyna P, Namenek Brouwer RJ, Fish LJ, Myers ER. Challenges and solutions for recruiting pregnant smokers into a nicotine replacement therapy trial. Nicotine Tob Res. 2006 Aug;8(4):547-54. doi: 10.1080/14622200600789882. PMID 16920652
- [Background] Bursey-Reddick, K, Swamy, GK, Brouwer, RN, Pollak, KI, Myers, ER. (2006). Comparison of Self-Reported Smoking Status and Anonymous Urinary Cotinine Testing in Pregnancy. American Journal of Obstetrics & Gynecology, 193 Supplement 6:S107.
- [Result] Pollak KI, Oncken CA, Lipkus IM, Lyna P, Swamy GK, Pletsch PK, Peterson BL, Heine RP, Brouwer RJ, Fish L, Myers ER. Nicotine replacement and behavioral therapy for smoking cessation in pregnancy. Am J Prev Med. 2007 Oct;33(4):297-305. doi: 10.1016/j.amepre.2007.05.006. PMID 17888856
- [Derived] Swamy GK, Roelands JJ, Peterson BL, Fish LJ, Oncken CA, Pletsch PK, Myers ER, Whitecar PW, Pollak KI. Predictors of adverse events among pregnant smokers exposed in a nicotine replacement therapy trial. Am J Obstet Gynecol. 2009 Oct;201(4):354.e1-7. doi: 10.1016/j.ajog.2009.06.006. Epub 2009 Aug 7. PMID 19664750